CLINICAL TRIAL: NCT06707363
Title: Psychological Predictors of Pain Experience in Patients After Emergency and Elective Orthopedic Surgery: a Longitudinal Study
Brief Title: Psychological Factors and Pain in Orthopedic Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Collaborators: Stefan Żeromski Specialist Hospital, Kraków (Unknown)
Responsible Party: Principal Investigator, Katarzyna Brzezewska, Principal Investigator, Psychologist, Jagiellonian University
Other Study IDs: KE/3_2023
Record Dates: First submitted 2024-11-12; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Orthopedic Surgical Procedures
Keywords: body image; emotional regulation; dysfunctional personality traits; pain experience; orthopedic surgery; subjective pain intensity
MeSH Terms: conditions — Emotional Regulation | interventions — Orthopedic Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- After orthopedic surgeries: This study focuses on patients who have undergone either emergency or elective orthopedic surgeries, specifically those involving significant interventions on the musculoskeletal system, such as joint replacements or fracture repairs. The cohort consists of adult participants (aged 18 years and older) who have been informed about the study and provided their consent to participate. This population will include both males and females.
  Interventions of interest: psychological questionnaires, pain assessment, longitudinal follow-up.
  Interventions: Procedure: orthopedic surgery

INTERVENTIONS:
Procedure: orthopedic surgery — Surgeries involving major interventions on the musculoskeletal system, such as joint replacement surgeries or fracture repairs.

SUMMARY:
The goal of this observational study is to verify the association of previously underexplored psychological variables on postoperative pain experience and its progression over time in patients undergoing emergency and elective orthopedic surgeries, including both sexes (age range: 18-65). The main questions it aims to answer are:

1. Do psychological factors such as dysfunctional personality traits and emotional regulation explain the experience of pain after surgery and after six months?
2. Does the experience of the body mediate the relationship between dysfunctional personality traits and the experience of pain after surgery and after six months?
3. Does the experience of pain differ between patients who underwent emergency and elective orthopedic surgery (after surgery and after six months)?

Researchers will compare the pain experience of patients undergoing emergency orthopedic surgery to those undergoing elective orthopedic surgery to see if there are significant differences in pain outcomes and recovery trajectories.

Participants will:

* complete psychological questionnairs to evaluate dysfunctional personality traits, emotional regulation, and body image;
* report their subjective pain level and provide information on their coping strategies for managing pain and information about pain interference in everyday functioning;
* engage in follow-up evaluation (6 months after the surgery) to assess the impact of pain on their daily activities and rehabilitation progress and complete some of the questionnaires again.

DETAILED DESCRIPTION:
The primary goal of the project is to formulate empirically grounded theses on the association of psychological variables and the type of pain experienced preoperatively on shaping the pain experience among orthopedic patients. Psychological variables, selected based on the literature, include dysfunctional personality traits, emotional regulation, and body image, while the pain experience is understood as the subjective level of pain experienced, pain coping strategies, and pain interference in daily functioning. Additionally, the project aims to compare the pain experience of patients undergoing emergency versus elective orthopedic surgeries in a longitudinal perspective, allowing for consideration of the dynamic nature of pain and its development over time. Orthopedic surgeries are considered among the most painful as they involve significant intervention in both the skeletal system and surrounding soft tissues. Postoperative discomfort often extends beyond acute pain, with 19-22% of orthopedic patients developing chronic pain after surgery. Many orthopedic patients experience reduced mobility and require rehabilitation-their pain experience and associated challenges may be unique. Furthermore, orthopedic surgery is invasive and deeply impacts body boundaries. Therefore, the study also seeks to examine the role of body image (as a mediating variable) in shaping the pain experience.

The research questions addressed will provide recommendations for pain management that highlight the importance of a biopsychosocial perspective, as well as recommendations for developing preventive and therapeutic programs for psychological work with orthopedic patients based on the study's findings.

Plan of the project Phase 1 - Data Collection: This will take place at the Department of Orthopedic and Traumatic Surgery of Żeromski Hospital in Krakow. Physicians will identify eligible patients based on inclusion and exclusion criteria, after which the researcher will seek patient consent for participation. A total of 170 patients aged 18-65 years who underwent elective or emergency orthopedic surgery will participate, completing questionnaires within 72 hours post-surgery. The following tools will be used: The Personality Inventory for ICD-11 (PiCD), Difficulties in Emotion Regulation Scale (DERS), The Pain Coping Strategies Questionnaire (CSQ), Visual analogue scale (VAS), Multidimensional Body Self Relations Questionnaire (MBSRQ), and Pain Interference Scale. Relevant medical information will be collected to control for confounding variables. This phase aims to generate empirical data on selected psychological variables and postoperative pain characteristics.

Phase 2 - Follow-up: This will occur six months postoperatively via online questionnaires, where patients will complete some of the previous questionnaires again. This phase aims to collect empirical data to (1) analyze changes in the pain experience over time and (2) analyze changes in body image and pain coping strategies over time post-surgery.

Data Analysis: Analysis of empirical data in SPSS will include mediation analysis, stepwise regression analysis, and analysis of group mean differences. This will support the following research objectives: (1) identification of psychological variables explaining postoperative pain experience and its changes over time; (2) comparative analysis of pain experiences among emergency versus elective surgery patients; (3) identification of the role of body image as a mediator between psychological variables and pain experience.

Interpretation of Results: Formulating conclusions from the analyses to achieve the main research objective: to empirically establish theses on (a) the impact of psychological variables; and (b) the impact of the type of pain experienced preoperatively on shaping the pain experience among orthopedic patients.

Dissemination of Results: Preparing study results in the form of articles, conference presentations, and popularization efforts to achieve the following research objectives: (1) providing recommendations for pain management that emphasize the need to consider a biopsychosocial perspective, particularly for orthopedic patients; (2) providing recommendations for developing preventive and therapeutic programs for psychological work with orthopedic patients based on the study's findings.

ELIGIBILITY:
Inclusion Criteria:

* age: participants aged 18 years or older;
* surgical procedures: individuals scheduled to undergo either emergency or elective orthopedic surgeries, including but not limited to joint replacements (e.g., hip or knee arthroplasty) and fracture repairs;
* time after operation: undergoing orthopedic surgery up to 72 hours before the psychological examination;
* informed consent: ability to provide informed consent and willingness to participate in the study;
* language proficiency: proficiency in the language of the questionnaires used in the study (Polish).

Exclusion Criteria:

* psychiatric disorders: diagnosed psychiatric disorders (e.g., severe depression, anxiety disorders) that are not managed or stable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on patients who have undergone either emergency or elective orthopedic surgeries, specifically those involving significant interventions on the musculoskeletal system, such as joint replacements or fracture repairs. The source of study participants is Stefan Żeromski Specialist Hospital in Krakow, Department of Orthopedic and Trauma Surgery.
  The cohort consists of adult participants (aged 18 years and older) who have been informed about the study and provided their consent to participate. This population will include both males and females. Interventions of interest: psychological questionnaires, pain assessment, longitudinal follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Dysfunctional personality traits | from 24 to 72 hours after surgery
  Variable defined as a set of traits describing an excessive (non-adaptive to maintaining health) intensity of basic personality traits. This variable consists of the following components: anankastia, disinhibition, negative affectivity, dissociality, and social isolation.
  Measurement Tool: The Personality Inventory for ICD-11 (PiCD). The PiCD includes items scored on a Likert scale from 1 to 5, where:
  1 indicates the lowest presence of a given trait. 5 indicates the highest presence of a given trait. Higher scores represent a greater intensity of dysfunctional personality traits, reflecting a non-adaptive psychological profile that may influence postoperative outcomes. Maximum possible score is 300.
Body image after surgery | from 24 to 72 hours after surgery
  Variable defined as a multidimensional construct that includes subjective thoughts, beliefs, feelings, and behaviors related to the body and physical functioning of the individual.
  Measurement Tool: The Multidimensional Body Self Relations Questionnaire (MBSRQ). This questionnaire consists of multiple subscales, each scored on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
  The minimum score on each subscale indicates a lower level of body image satisfaction or awareness.
  The maximum score indicates a higher level of body image satisfaction or awareness. The maximum possible score is 345.
Emotion regulation after sugery | from 24 to 72 hours after surgery
  Refers to challenges in the process of modulating emotions to facilitate the achievement of specific goals.
  Measurement Tool: The Difficulties in Emotion Regulation Scale (DERS). This scale measures various aspects of emotion regulation difficulties across multiple subscales.
  Scores on each subscale range from 1 (indicating fewer difficulties) to 5 (indicating greater difficulties).
  Minimum total score: reflects lower levels of emotion regulation difficulties. Maximum total score: indicates higher levels of difficulties in regulating emotions. Maximum possible score is 180.
Subjective pain severity after surgery | from 24 to 72 hours after surgery
  Subjective pain severity measured by Visual analogue scale (VAS). It takes the form of a horizontal line of 10 centimeters long. The patient draws a vertical line on it indicating the intensity of the pain from 0 (no pain at all) to 10 (worst pain imaginable).
Pain coping strategies after surgery | from 24 to 72 hours after surgery
  Understood as taking action to minimize pain, reduce its impact on daily functioning, and alleviate emotional tension caused by pain.
  Measurement Tool: The Pain Coping Strategies Questionnaire (CSQ). This questionnaire assesses the frequency and type of coping strategies used by individuals to manage pain.
  Scores on individual strategies range from 0 (indicating no use of a specific strategy) to 6 (indicating frequent use).
  Minimum total score: indicates less use of pain-coping strategies. Maximum total score: reflects greater reliance on coping strategies. Higher scores in adaptive coping strategies (e.g., distraction, cognitive reinterpretation) suggest better pain management outcomes, while higher scores in maladaptive strategies (e.g., catastrophizing) indicate worse outcomes. Maximum possible score is 252.
Pain interference with daily functioning (after surgery) | from 24 to 72 hours after surgery
  Defined as the level at which pain disrupts daily functioning. Pain interference is measured by 11 questions addressing various areas of life, including rest, physical fitness, mood, household and professional duties, relationships with others, intellectual activities, and sexual activity.
  Scale: Each question is rated on a 5-point Likert scale (1 = no interference, 5 = extreme interference). Minimum total score: indicates minimal disruption caused by pain. Maximum total score: reflects severe interference in all assessed areas. Higher scores in specific subscales (e.g., mood, physical fitness) suggest greater pain-related challenges in those domains. Maximum possible score is 55.
Socialdemographic and medical data | from 24 to 72 hours after surgery
  Information such as age, sex, education, occupation, marital status, type of orthopedic surgery, surgical anesthesia, painkillers taken, chronic diseases, previous surgeries, rehabilitation undertaken.

SECONDARY OUTCOMES:
Body image (6 months later) | 6 months after surgery
  Variable defined as a multidimensional construct that includes subjective thoughts, beliefs, feelings, and behaviors related to the body and physical functioning of the individual. Measurement Tool: The Multidimensional Body Self Relations Questionnaire (MBSRQ). This questionnaire consists of multiple subscales, each scored on a Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The minimum score on each subscale indicates a lower level of body image satisfaction or awareness. The maximum score indicates a higher level of body image satisfaction or awareness. The maximum possible score is 345.
Emotion regulation (6 months after surgery) | 6 months after surgery
  Refers to challenges in the process of modulating emotions to facilitate the achievement of specific goals. Measurement Tool: The Difficulties in Emotion Regulation Scale (DERS). This scale measures various aspects of emotion regulation difficulties across multiple subscales. Scores on each subscale range from 1 (indicating fewer difficulties) to 5 (indicating greater difficulties). Minimum total score: reflects lower levels of emotion regulation difficulties. Maximum total score: indicates higher levels of difficulties in regulating emotions. Maximum possible score is 180.
Subjective pain severity (6 months after surgery) | 6 months after surgery
  Subjective pain severity measured by Visual analogue scale (VAS). It takes the form of a horizontal line of 10 centimeters long. The patient draws a vertical line on it indicating the intensity of the pain from 0 (no pain at all) to 10 (worst pain imaginable).
Pain coping strategies (6 months after surgery) | 6 months after surgery
  Understood as taking action to minimize pain, reduce its impact on daily functioning, and alleviate emotional tension caused by pain. Measurement Tool: The Pain Coping Strategies Questionnaire (CSQ). This questionnaire assesses the frequency and type of coping strategies used by individuals to manage pain. Scores on individual strategies range from 0 (indicating no use of a specific strategy) to 6 (indicating frequent use). Minimum total score: indicates less use of pain-coping strategies. Maximum total score: reflects greater reliance on coping strategies. Higher scores in adaptive coping strategies (e.g., distraction, cognitive reinterpretation) suggest better pain management outcomes, while higher scores in maladaptive strategies (e.g., catastrophizing) indicate worse outcomes. Maximum possible score is 252.
Pain interference with daily functioning (6 months after surgery) | 6 months after surgery
  Defined as the level at which pain disrupts daily functioning. Pain interference is measured by 11 questions addressing various areas of life, including rest, physical fitness, mood, household and professional duties, relationships with others, intellectual activities, and sexual activity. Scale: Each question is rated on a 5-point Likert scale (1 = no interference, 5 = extreme interference). Minimum total score: indicates minimal disruption caused by pain. Maximum total score: reflects severe interference in all assessed areas. Higher scores in specific subscales (e.g., mood, physical fitness) suggest greater pain-related challenges in those domains. Maximum possible score is 55.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadetta Izydorczyk, Psychology Professor, Study Director — Jagiellonian University
Locations (2):
- Poland (2):
  - Stefan Żeromski Specialist Hospital in Krakow, Department of Orthopedic and Trauma Surgery, Krakow, Malopolska
  - Stefan Żeromski Specialist Hospital, Krakow, Malopolska

IPD SHARING:
Plan to Share IPD: Yes
* data dictionary (a description of the variables)
  * demographic data
  * outcome measures
Supporting Information: ICF
URL: https://uj.rodbuk.pl/

REFERENCES:
- [Background] Khan RS, Ahmed K, Blakeway E, Skapinakis P, Nihoyannopoulos L, Macleod K, Sevdalis N, Ashrafian H, Platt M, Darzi A, Athanasiou T. Catastrophizing: a predictive factor for postoperative pain. Am J Surg. 2011 Jan;201(1):122-31. doi: 10.1016/j.amjsurg.2010.02.007. Epub 2010 Sep 15. PMID 20832052
- [Background] Khalil H, Shajrawi A, Dweik G, Zaghmouri A, Henker R. The impact of preoperative pain-related psychological factors on pain intensity post-surgery in Jordan. J Health Psychol. 2021 Dec;26(14):2876-2885. doi: 10.1177/1359105320937067. Epub 2020 Jun 27. PMID 32597221
- [Background] Correll D. Chronic postoperative pain: recent findings in understanding and management. F1000Res. 2017 Jul 4;6:1054. doi: 10.12688/f1000research.11101.1. eCollection 2017. PMID 28713565
- [Background] Burns LC, Ritvo SE, Ferguson MK, Clarke H, Seltzer Z, Katz J. Pain catastrophizing as a risk factor for chronic pain after total knee arthroplasty: a systematic review. J Pain Res. 2015 Jan 5;8:21-32. doi: 10.2147/JPR.S64730. eCollection 2015. PMID 25609995